CLINICAL TRIAL: NCT01931553
Title: Back to Bedside: A Pragmatic Cluster Randomized Controlled Trial to Standardize Attending Morning Rounds in Medicine
Brief Title: A Pragmatic Cluster Randomized Controlled Trial to Standardize Attending Morning Rounds in Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: RoundingUCSF
Record Dates: First submitted 2013-08-16; First posted 2013-08-29 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Morning Rounds; Teaching Rounds; Hospitalization; Inpatients; Quality Improvement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standardized attending morning rounds (Experimental): 1. Pre-rounds discretion
  2. Pre-rounds huddle
  3. Bedside RN integration
  4. Patient-centered rounding
  5. Real-time order writing
  Interventions: Other: Standardized attending morning rounds
- Usual rounding practice (No Intervention): Usual rounding practice (as defined by each clinical team)

INTERVENTIONS:
Other: Standardized attending morning rounds
  Arms: Standardized attending morning rounds

SUMMARY:
Attending morning rounds take place at teaching hospitals every day. They are the primary mechanism for patient care delivery, supervision and education of trainees, and communication with patients, families, and staff. However, they are done with little standardization or widely recognized best practices.

The objective of this quality improvement (QI) initiative is to evaluate the adherence to and impact of implementing standardized attending morning rounds on medicine teams at our institution. A standardized rounding intervention has been developed which includes specific guidance on completing the following activities during morning rounds: (1) Pre-rounds discretion; (2) Pre-rounds huddle; (3) Bedside registered nurse (RN) integration; (4) Patient-centered rounding; (5) Real-time order writing.

This trial will randomize half of the investigators' medicine teams at University of California San Francisco to this rounding intervention whilst the other half will be randomized to continue with usual unstandardized rounding practices.

The investigators will compare medicine teams randomized to undertake standardized rounding to those teams undertaking usual practice. Outcomes assessed will relate to the patient (e.g. satisfaction), providers (e.g. satisfaction), efficiency (e.g. total morning round time) as well as adherence to the intervention .

The investigators' study hypotheses are that patient satisfaction scores will be higher for those patients receiving standardized bedside rounds compared to the usual care group. The investigators also hypothesize that total attending morning rounds time and interns length of workday will be shorter and that the number of consultations ordered before noon will increase for those teams undertaking standardized bedside. Further, the investigator hypothesize higher levels of nurse participation, physician and medical student satisfaction with standardized bedside rounding.

ELIGIBILITY:
Inclusion Criteria:

* All attending physicians, residents, interns and medical students of Medicine teams A through H
* All patients admitted to Medicine teams A through H
* All nurses on the Medicine floors

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with morning rounds | Once, after day one of hospitalization and before patient is discharged.
  Patient satisfaction with morning ward rounds. This inpatient assessment will occur after day one of hospitalization before the patient is discharged from hospital. This time point will ensure that patients have experienced rounds at least once before completing a patient satisfaction survey.
Patient satisfaction with provider communication | Once, within one month of hospital discharge
  Post-discharge assessment will be sent by a commercial Vendor (Press Ganey) within a month of discharge following hospitalization

SECONDARY OUTCOMES:
Interns total length of workday | Daily during the 3-month trial
  The interns total length of workday will be recorded daily. Over the course of the trial the average length of workday will be determined including any duty hour violations.
Number of consultations ordered before noon | Daily during the 3-month trial
  The number of consultations ordered before noon will be recorded daily. Over the course of the trial the average number of consultations ordered before noon will be calculated.
Resident satisfaction | Once during the last week of their rotation on a given team
  Resident satisfaction and perceptions of with morning rounds (e.g. efficiency, organization, educational value)
Attending physician satisfaction | Once during the last week of their rotation on a given team
  Attending physician satisfaction and perceptions of with morning rounds (e.g. efficiency, organization, educational value)
Medical student satisfaction | Once during the last week of their rotation on a given team
  Medical student satisfaction and perceptions of with morning rounds (e.g. efficiency, organization, educational value)
Nurse participation in morning rounds | Daily during the 3-month trial
  The presence of RN during morning ward rounds will be recorded daily.
Nurse satisfaction | Once during the last week the trial
  Nurse satisfaction and perceptions of with morning rounds (e.g. efficiency, organization, team work)
Intern satisfaction | Once during the last week of their rotation on a given team
  Intern satisfaction and perceptions of with morning rounds (e.g. efficiency, organization, educational value)
Total morning rounding time | Daily during the 3-month trial
  Total morning rounding time will be recorded daily for each team. Over the course of the trial the average length of morning rounds will be determined.

OTHER OUTCOMES:
Number of discharges before noon | Daily during the 3-month trial
Cost of care per patient | For entire 3 month study period
  Average cost of care per patients for each group for entire 3-month study period
Length of stay | For entire 3 month study period
  Average length of stay for each group for entire 3-month study period
30-day readmission rate | For entire 3 month study period
  Average readmission rate for each group for entire 3-month study period
Adherence to the intervention | Daily during the 3-month trial
  Adherence to the standardized intervention will be recorded throughout the trial to determine the uptake of this intervention in everyday practice.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Monash, MD, Principal Investigator — University of California, San Francisco; Nader Najafi, MD, Principal Investigator — University of California, San Francisco; James D Harrison, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Monash B, Najafi N, Mourad M, Rajkomar A, Ranji SR, Fang MC, Glass M, Milev D, Ding Y, Shen A, Sharpe BA, Harrison JD. Standardized Attending Rounds to Improve the Patient Experience: A Pragmatic Cluster Randomized Controlled Trial. J Hosp Med. 2017 Mar;12(3):143-149. doi: 10.12788/jhm.2694. PMID 28272589